CLINICAL TRIAL: NCT04187534
Title: Critical Care Optimization of Albumin Ordering
Acronym: RATIONALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Daniel Niven, Assistant Professor, University of Calgary
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-1143
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Critical Illness
Keywords: Albumin; fluid resuscitation; de-adoption; de-implementation; low-value care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Registry-based, stepped-wedge, implementation trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin Fluid Resuscitation Optimization Intervention (Experimental): Our quality improvement intervention seeking to improve appropriate use and reduce inappropriate use of albumin for fluid resuscitation will consist of establishing a clinical champion, educating clinicians, changing the process for albumin ordering through development of an albumin order sheet, and providing quarterly unit-level audit/feedback data to clinicians on albumin utilization.
  Interventions: Other: Albumin Fluid Resuscitation Optimization Intervention
- Usual Practice (Active Comparator): Stepped-wedge roll out of 'Albumin Fluid Resuscitation Optimization Intervention' will permit those ICUs wherein intervention has not yet been implemented to serve as controls. These ICUs will prescribe albumin according to usual practice and not be exposed to any components of the intervention.
  Interventions: Other: Usual Practice

INTERVENTIONS:
Other: Albumin Fluid Resuscitation Optimization Intervention — Multi-faceted quality improvement intervention to optimize appropriateness of albumin use for fluid resuscitation
  Arms: Albumin Fluid Resuscitation Optimization Intervention
Other: Usual Practice — Albumin fluid resuscitation according to usual practice
  Arms: Usual Practice

SUMMARY:
Strong evidence suggests that human albumin solutions should not be used for fluid resuscitation except among patients undergoing therapeutic plasmapheresis and select patients with complications of liver cirrhosis (i.e. spontaneous bacterial peritonitis, or large volume ascitic fluid removal). Previous work by the investigators reported albumin use outside these circumstances as a quality improvement opportunity in Alberta ICUs. In 2017, the investigators began a pilot initiative to reduce albumin overuse in 6 ICUs in Alberta. The intervention was developed according to the Theoretical Domains Framework, and consisted of establishing a clinical champion, educating clinicians, changing the process for albumin ordering (albumin-specific order sheet), and providing quarterly audit/feedback data to clinicians on albumin utilization. During the intervention, there was a 41% relative reduction in albumin utilization. However, follow-up data identified problems with sustainability. These sustainability challenges combined with data suggesting high albumin use in other ICUs throughout Alberta have led the current project to build on the pilot initiative to reduce albumin overuse within all adult ICUs in Alberta.

The proposed quality improvement intervention will be implemented in 16 adult ICUs using a registry-based, stepped-wedge implementation design that will lean heavily on existing Provincial healthcare infrastructure. The intervention was developed using the Theoretical Domains Framework, and tailored to the unique features of each participating ICU. It will be implemented at the level of ICU. Clusters of 2 ICUs will be assigned to receive the intervention every month such that all ICUs in Alberta will receive the intervention by the end of the implementation period. To evaluate the quality improvement initiative, eCritical will serve as a 'registry' and will be used to capture all clinical and outcome data. The primary outcome will be the proportion of ICU admissions without an evidence-based indication for albumin, prescribed at least 1 unit of albumin (any concentration) during admission to ICU. 'Evidence-based indication' will be operationally defined as receipt of therapeutic plasmapheresis OR having a diagnosis of liver cirrhosis and being in receipt of a paracentesis. This latter criterion enables identification of patients with spontaneous bacterial peritonitis or large volume ascitic fluid removal.

DETAILED DESCRIPTION:
BACKGROUND: Strong evidence suggests that human albumin solutions should not be used for fluid resuscitation except among patients undergoing therapeutic plasmapheresis and select patients with complications of liver cirrhosis (i.e. spontaneous bacterial peritonitis, or large volume ascitic fluid removal). Previous work by the investigators reported overuse of albumin fluid resuscitation as a stakeholder-identified quality improvement opportunity in Alberta ICUs. Audit data from the provincial electronic medical record (EMR) for critical care, eCritical, reinforced stakeholder opinion and demonstrated that within Alberta ICUs in 2016 a considerable amount of albumin use deviated from evidence-based indications. On average, 14% of admissions to adult ICUs received at least one albumin unit during their ICU admission, with several high-use units providing albumin to between 20% and 35% of admissions. In 2017 the investigators began a pilot quality improvement initiative to reduce albumin overuse in six ICUs in Alberta. The intervention was developed according to the Theoretical Domains Framework. Questionnaires completed by clinicians working in the target ICU identified local culture and opinion of clinical leaders as barriers, and education, order sets, and clinical champions as facilitators to reducing albumin use. The intervention thus consisted of establishing a clinical champion, educating clinicians, changing the process for albumin through development of an albumin order sheet, and providing quarterly unit-level audit/feedback data to clinicians on albumin utilization. There was a 41% reduction in albumin utilization, however follow-up data identified problems with sustainability. The current project will build on the pilot initiative to implement a quality improvement intervention to reduce albumin overuse within all adult ICUs in Alberta.

OBJECTIVE: Evaluate albumin reduction within all adult ICUs in Alberta.

METHODS: This will be a registry-based, stepped-wedge quality improvement initiative.

Quality Improvement Initiative: Spread to 16 adult ICUs in Alberta will require understanding and adapting the investigators pilot intervention to local barriers and facilitators. The intervention for this quality improvement initiative will be developed using the Theoretical Domains Framework. The research team will develop working groups responsible for tailoring the intervention and implementation strategy to each participating ICU. This will be conducted as part of the Province-wide quality improvement initiative. The investigators will conduct the quality improvement initiative using a registry-based, stepped-wedge, implementation trial. Owing to the nature of this design, the interventions will be implemented at the level of ICU. Clusters of 2 ICUs will be assigned to receive the intervention every month such that all ICUs in Alberta will receive the intervention by the end of the implementation period.

Registry-based data analysis: To evaluate this quality improvement initiative, the Provincial EMR for critical care, eCritical, will serve as a 'registry' and will be used to capture all clinical and outcome data. Data will be collected until patient death or hospital discharge and censored at 60 days. To optimize efficiency and power, data will be collected 3-months before and after implementation of the interventions.

SETTING: 16 adult ICUs in Alberta's critical care strategic clinical network reflecting teaching/non-teaching and urban/rural hospitals will participate.

STUDY POPULATION: All adult patients (>18 years) admitted to the study ICUs during the study period (November 2019 to January 2021). Study ICUs will include 14 general medical-surgical ICUs, and 2 cardiovascular surgery ICUs.

OUTCOMES: The primary outcome of this study will be the proportion of ICU patients without an evidence-based indication for albumin prescribed at least 1 unit of albumin (any concentration) during admission to ICU. Evidence-based indication will be operationally defined as receipt of therapeutic plasmapheresis OR having a diagnosis of liver cirrhosis and being in receipt of a paracentesis. This latter criterion enables identification of patients with either spontaneous bacterial peritonitis or large volume ascitic fluid removal. This outcome was selected because: 1) there is precedent within current literature; 2) previous experience auditing albumin utilization in Alberta ICUs demonstrate it is available through eCritical; 3) it provides a relevant, broadly understandable estimate of the effect of the implementation science intervention to change albumin overuse; and 4) it permits assessment of the feasibility of implementing the platform to develop and carry out multi-stakeholder implementation science interventions to promote evidence-informed clinical practices and evaluate the intervention.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the study ICUs

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50000 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of ICU admissions receiving albumin | During ICU admission
  Proportion of ICU admissions without an evidence-based indication for albumin prescribed at least 1 unit of albumin (any concentration) during admission to ICU

SECONDARY OUTCOMES:
Mean number of albumin units among those receiving albumin | During ICU admission
  Mean number of albumin units prescribed to patients without an evidence-based indication for albumin that received at least 1 unit of albumin
Total fluid administration | ICU day 7
  Total volume of fluid administered during days 1-7 in ICU
Total crystalloid fluid | ICU Day 7
  Total volume of crystalloid fluid administered during days 1-7 in ICU
Duration of vasopressor administration | From date of ICU admission to date of discharge, on average 1-6 days
  Number of days vasopressors administered during ICU length of stay
Length of mechanical ventilation | From date mechanical ventilation commended to date discontinued, on average 0-3 days
  Number of days on mechanical ventilation from time of starting mechanical ventilation during ICU length of stay
ICU length of stay | From date of ICU admission to date of discharge, on average 1-6 days
  Number of days admitted to ICU (unique number per admission)
Hospital length of stay | From date of hospital admission to date of discharge, on average 5-20 days
  Number of days admitted to hospital (unique number per admission)
ICU mortality | From date of ICU admission to date of discharge, on average 1-6 days
  Survival to discharge from ICU
Hospital mortality | From date of hospital admission to date of discharge, on average 5-20 days
  Survival to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Niven, MD, PhD, Principal Investigator — University of Calgary
Locations (15):
- Canada (15):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Mazankowski Heart Institute, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nun's Hospital, Edmonton, Alberta
  - Northern Lights Regional Health Centre, Fort McMurray, Alberta
  - Queen Elizabeth II Hospital, Grande Prairie, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - Red Deer Regional Hospital Centre, Red Deer, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sauro K, Bagshaw SM, Niven D, Soo A, Brundin-Mather R, Parsons Leigh J, Cook DJ, Stelfox HT. Barriers and facilitators to adopting high value practices and de-adopting low value practices in Canadian intensive care units: a multimethod study. BMJ Open. 2019 Mar 15;9(3):e024159. doi: 10.1136/bmjopen-2018-024159. PMID 30878979